CLINICAL TRIAL: NCT06712875
Title: A Pilot Study Evaluating the Toxicity and Clinical Benefit of Mitogen-activated Protein Kinase (MAPK) Pathway Inhibition Combined With Programmed Cell Death-1 Checkpoint Blockade (Anti-PD1) for the Treatment of BRAF-altered Pediatric Gliomas
Brief Title: MAPK Inhibition Combined With Anti-PD1 Therapy for BRAF-altered Pediatric Gliomas
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Ashley S. Plant, MD, Principal Investigator, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCH24C02
Record Dates: First submitted 2024-11-26; First posted 2024-12-02 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Low Grade Glioma; High Grade Glioma
Keywords: BRAF; BRAFV600; KIAA1549 BRAF fusion; nivolumab; dabrafenib; trametinib; MAPK inhibition combined with anti-PD1 immunotherapy; recurrent low grade glioma; high grade glioma
MeSH Terms: conditions — Glioma | interventions — trametinib; Nivolumab; dabrafenib

STUDY DESIGN:
Intervention Model Description: Pilot study evaluating toxicity and early efficacy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Trametinib combined with nivolumab (Cohort A) (Experimental): Patients with histologically confirmed diagnosis of pediatric high- or low-grade glioma harboring a KIAA1549-BRAF fusion. Patients with NF1-associated gliomas or NF1-altered glioma.
  Patients in Cohort A will receive trametinib and nivolumab combination therapy. Trametinib will be administered at 0.025 mg/kg/dose orally once daily.
  Nivolumab will be administered at 6 mg/kg/dose intravenously every 4 weeks.
  Cycle length will be every 28 days. Treatment will include 1 year or 13 cycles of combination therapy, whichever comes first. For patients with high grade glioma, therapy can be continued beyond the 13 cycles if they are deemed to have clinical benefit from the therapy. Patients will be followed for up to 5 years to evaluate clinical endpoints.
  Interventions: Drug: Trametinib and Nivolumab
- Dabrafenib + trametinib combined with nivolumab (Cohort B) (Experimental): Patients with histologically confirmed diagnosis of pediatric low-grade glioma harboring a BRAFV600 mutation that is recurrent or progressive or non-brainstem pediatric high-grade glioma harbor ng BRAFV600 mutation that is newly diagnosed, recurrent, or progressive.
  Cohort B will receive trametinib, nivolumab dabrafenib combination therapy. Trametinib will be administered at 0.025 mg/kg/dose orally once daily.
  Nivolumab will be administered at 6 mg/kg/dose intravenously every 4 weeks. Dabrafenib will be administered at a dose of 5.25 mg/kg/day orally divided into two doses, which shall be taken 12 hours apart.
  Cycle length will be every 28 days. Treatment will include 1 year or 13 cycles of combination therapy, whichever comes first. For patients with high grade glioma, therapy can be continued beyond the 13 cycles if they are deemed to have clinical benefit from the therapy. Patients will be followed for up to 5 years to evaluate clinical endpoints.
  Interventions: Drug: Dabrafenib, trametinib, nivolumab

INTERVENTIONS:
Drug: Trametinib and Nivolumab — Trametinib combined with nivolumab (Cohort A)
  Arms: Trametinib combined with nivolumab (Cohort A)
Drug: Dabrafenib, trametinib, nivolumab — Dabrafenib + trametinib combined with nivolumab (Cohort B)
  Arms: Dabrafenib + trametinib combined with nivolumab (Cohort B)

SUMMARY:
Pediatric gliomas harboring BRAF-alterations, commonly BRAFV600 mutation or KIAA1549-BRAF fusion, are currently treated with either chemotherapy or mitogen activated protein kinase (MAPK) inhibitors, such as, dabrafenib and/or trametinib. Unfortunately, some BRAF-altered gliomas can progress or have rebound growth after discontinuation of therapy. Data from BRAFV600E-mutant melanoma has shown potential synergy between MAPK inhibition and anti-programmed cell death 1 (anti-PD1) checkpoint blockade. Anti-PD1 therapy, such as, nivolumab can block the PD1 receptor on T cells, a marker of T cell exhaustion, allowing a continued or more robust anti-tumor immune response. Here, investigators will combine MAPK inhibition with anti-PD1 therapy in recurrent, refractory low grade BRAF-altered glioma and newly diagnosed or recurrent BRAF-altered or NF-altered high grade glioma.

DETAILED DESCRIPTION:
This is a pilot study evaluating the toxicity and early efficacy of dabrafenib and/or trametinib combined with nivolumab for the treatment of BRAF-altered or NF altered gliomas. While dabrafenib, trametinib, and nivolumab have been used for pediatric gliomas in previous studies, this will be the first pediatric study evaluating the combination of these agents.

This study will evaluate the use of dabrafenib, trametinib, and nivolumab in patients in recurrent, refractory, or progressive low grade gliomas harboring BRAFV600 mutations who have previously been treated with MAPK inhibition alone. The same combination will be explored in newly diagnosed or recurrent BRAFV600 mutant high grade glioma.

This study will also evaluate the use of trametinib and nivolumab in patients with recurrent, refractory, or progressive low grade gliomas harboring a KIAA1549 BRAF fusion who have previously been treated with MAPK inhibition alone. The same combination will be explored in NF altered transforming or high grade glioma or high grade glioma harboring a KIAA1549 BRAF fusion.

The objective of this study is to understand the safety and tolerability of the combination of dabrafenib, trametinib, and/or nivolumab in pediatrics. Secondarily, this study will evaluate for an early efficacy signal of the combination therapy and compare to historical treatment response to MAPK inhibition alone.

ELIGIBILITY:
Inclusion Criteria:

Cohort A Only:

* Patients with histologically confirmed diagnosis of pediatric high- or low-grade glioma harboring a KIAA1549-BRAF fusion: Low-grade glioma that is recurrent or progressive OR High-grade glioma that is newly diagnosed or recurrent OR
* Patients with NF1-associated gliomas or NF1-altered glioma: Low-grade glioma that is recurrent or progressive OR High-grade glioma that is newly diagnosed or recurrent OR Transforming glioma that is newly diagnosed or recurrent

Cohort B Only:

* Patients with histologically confirmed diagnosis of pediatric low-grade glioma harboring a BRAFV600 mutation that is recurrent or progressive OR
* Patients with histologically confirmed diagnosis of non-brainstem pediatric high-grade glioma harboring BRAFV600 mutation that is newly diagnosed, recurrent, or progressive

All Cohorts:

* Patients must be ≥1 and ≤26 years of age at the time of enrollment.
* Patients must have a performance status of Karnofsky >50% for patients >16 years old and Lansky >50% for patients <16 years old.
* Patients must have adequate organ and bone marrow function
* The effects of dabrafenib, trametinib, and nivolumab on the developing human fetus are unknown. For this reason, patients of childbearing potential (POCBP) and patients with sperm-producing reproductive capacity (PWSPRC) must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) from time of informed consent for the duration of study participation and for 30 days following completion of therapy. POCBP must have a negative pregnancy test.
* Patients with neurological deficits that are stable for a minimum of 1 week prior to enrollment are eligible.

Note: A baseline detailed neurological exam should clearly document the neurological status of the patient at the time of enrollment on the study.

- Patients who are receiving dexamethasone must be on a stable or decreasing dose for at least 1 week prior to enrollment. Total dexamethasone dose at time of enrollment must be less than or equal to 2 mg/day total or 0.5 mg/kg/day, whichever is smaller.

LGG Only

* Patients must have received a prior BRAF inhibitor (first or second generation), MEK inhibitor, or a combination. The response to this therapy must be known and information provided at study enrollment.
* Patients must have recovered from acute treatment-related toxicities (defined as <Grade 1, excludes alopecia) prior to entering this study.

HGG Only

* Patients must have received prior radiotherapy >12 weeks prior to enrollment.
* Patients must have recovered from acute treatment-related toxicities (defined as <Grade 1, excludes alopecia) prior to entering this study.
* NF1 patients with transforming gliomas and high-grade gliomas are eligible regardless of prior systemic therapy.
* Patients who have received prior radiation therapy must have experienced progression post-radiation OR have measurable disease defined as residual tumor >1cm in at least one dimension

Exclusion Criteria:

* Patients with disseminated disease.
* Patients who have had prior radiation therapy <12 weeks prior to registration.
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 1) (with the exception of alopecia).
* Patients who receiving any other investigational agents. Note: There will be a 21-day washout period for all chemotherapeutic agents, a washout period of two half-lives for any targeted agents (e.g., MAPK inhibitors), and/or a washout period of 4 weeks for any antibody therapies (e.g., bevacizumab).
* Patients who have a history of allergic reactions attributed to compounds of similar chemical or biological composition to dabrafenib, trametinib, or nivolumab.
* Patients who have received MAPK inhibitor and checkpoint blockade combination therapy.

Note: Patients may have received MAPK inhibitor monotherapy or checkpoint blockade monotherapy.

* Patients who previously discontinued BRAF inhibitor (type 1 inhibitor or dimer inhibitor, such as, DAY101), MEK inhibitor, or the combination because of grade 3 or higher toxicity or clinically significant grade 2 toxicity requiring discontinuation of therapy are not eligible.
* Patients with the following:

  * Known autoimmune disorders
  * Immune disorders
  * Immunodeficiencies
* Patients with Crohn's disease, ulcerative colitis, or other inflammatory bowel disease.
* Patients with active pancreatitis or history of pancreatitis within the last 3 months.
* Patients with active interstitial lung disease (ILD)/pneumonitis or a history of ILD/pneumonitis requiring treatment with systemic steroids.
* Patients who have a known active Human Immunodeficiency Virus (HIV), Hepatitis B, or Hepatitis C infection are ineligible. Patient must have documented evidence of negative tests for the presence of HIV, Hepatitis B surface antigen, and Hepatitis C (anti-HCV antibody OR Hep C RNA-qualitative).
* Patients who have received a major surgical procedure ≤ 28 days of beginning study treatment, or minor surgical procedures (including VP shunt placement or stereotactic biopsy of the tumor) ≤ 7 days are not eligible.
* Patients who are taking herbal preparations. These medications include but are not limited to St. John's wort, kava, ephedra (ma hung), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, and ginseng. Cannabis products of any type are not allowed throughout the study. Patients should stop using these herbal medications or cannabis products 7 days prior to enrollment.
* Patients who are pregnant. Patients of childbearing potential must have a negative serum or urine pregnancy test. (If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.)
* Patients who are lactating (unless they have agreed to not breastfeed). Breastfeeding patients are excluded from this study due to risks of fetal and teratogenic adverse events as seen in animal/human studies.
* Patients with any clinically significant unrelated systemic illness (serious infections or significant cardiac, pulmonary, hepatic, or other organ dysfunction), that in the opinion of the investigator would compromise the patient's ability to tolerate protocol therapy, put them at additional risk for toxicity or would interfere with the study procedures or results.
* Patients with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen for this trial.
* Patients with bulky tumor on imaging are ineligible. Bulky tumor is defined as:

  * Tumor with any evidence of clinically significant uncal herniation or midline shift
  * Tumor with diameter of >5cm in one dimension on T2/FLAIR except for those patients with newly diagnosed HGG treated following irradiation without signs of tumor progression. For the latter group, a maximum diameter of contrast enhancing solid or necrotic tumor and of T2/FLAIR abnormality will be 5 cm and 8 cm, respectively.
  * Tumor that in the opinion of the site investigator, shows significant mass effect
  * Metastatic disease: Patients with ≤ 5 separate foci of metastatic disease not causing mass effect on adjacent parenchyma and each measuring less than 0.5 cm in maximum diameter will be eligible for this arm of the study. Patients with leptomeningeal disease are eligible.
  * Multi-focal disease (patients with multi-focal parenchymal disease will be eligible if the sum of the product of the maximum perpendicular diameters of all measurable non-contiguous lesions is less than 16 cm2 based on the T2/FLAIR abnormality).

Ages: 1 Year to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Safety based on number of participants with treatment-related adverse events based on scoring from CTCAE v4.0 | The dose limiting toxicity (DLT) period is 28 days.
  This study will utilize a rolling 6 design and enroll 12 evaluable patients in each cohort (Cohort A and B). Two dose levels will be utilized to assess safety and tolerability. Dose level 1 includes 100% dosing of dabrafenib and/or trametinib and nivolumab. A dose level -1 will be utilized if dose level 1 is not tolerable and will include 100% dosing of nivolumab with 70% dosing of dabrafenib and/or trametinib.

SECONDARY OUTCOMES:
Response assessment | From enrollment through end of treatment at 1 year
  Objective response rate will be utilized to assess response to combination therapy. Magnetic resonance imaging (MRI) will be evaluated for response utilizing RANO/iRANO criteria. Best response and duration of response be assessed. An objective response is a partial or complete response (PR or CR) sustained for at least 12 weeks.
Assessment of "Better Response" | From enrollment to the end of treatment at 1 year
  At enrollment, information will be entered by the study team regarding prior treatment with MAPK inhibition alone. The best response and duration of this response will be recorded. This will be compared to response on study treatment. A "better response" would be considered an improvement of best response from stable disease to partial response, partial response to complete response, or progressive disease to stable disease OR a similar best response that is maintained for 12 weeks longer or more.
Progression free survival | From enrollment through long term follow up (5 years post treatment)
  Progression will be determined by magnetic resonance imaging (MRI) assessment using RANO/iRANO criteria.
Overall Survival (OS) | Time of enrollment through long term follow up (5 years post treatment)
  Overall survival will be assessed by time to event (death).

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Plant-Fox, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (3):
- United States (3):
  - Children's National Hospital, Washington D.C., District of Columbia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: No
I do not plan to provide individual participant data except in de-identified format in publication or amongst study investigators